CLINICAL TRIAL: NCT00875901
Title: Hypofractionated, Image-Guided Radiation Therapy With Proton Therapy for Stage I Non-Small Cell Lung Cancer
Brief Title: Proton Therapy for Stage I Non-Small Cell Lung Cancer (LU03)
Acronym: LU03
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFPTI 0901 - LU03
Record Dates: First submitted 2009-04-02; First posted 2009-04-06 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Lung Cancer; Stage I Non-Small Cell Lung Cancer; Proton Radiation; HypoIGRT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peripherally located lung tumor (Experimental): 12 cobalt gray equivalent per fraction to a total of 48 cobalt gray equivalent
  Interventions: Radiation: Peripherally located lung tumor
- Centrally located lung tumor (Experimental): 6 cobalt gray equivalent per fraction to a total of 60 cobalt gray equivalent
  Interventions: Radiation: Centrally located lung tumor

INTERVENTIONS:
Radiation: Peripherally located lung tumor — 12 cobalt gray equivalent per fraction for 4 fractions, 2-3 treatments per week (every other day), over 2 weeks for a total of 48 cobalt gray equivalent (Fractions at lest 40 hours apart)
  Other Names: Proton Radiation
  Arms: Peripherally located lung tumor
Radiation: Centrally located lung tumor — 6 cobalt gray equivalent per fraction for 10 fractions, 5 treatments per week over 2-3 weeks for a total of 60 cobalt gray equivalent (no more than one fraction per calendar day)
  Other Names: Proton Radiation
  Arms: Centrally located lung tumor

SUMMARY:
This is a research study to determine if hypofractionated image guided radiation therapy (hypoIGRT) with proton therapy is a good way to treat early stage lung tumors for patients who will not have surgery. HypoIGRT delivers higher daily doses of radiation over a shorter period of time compared with conventional radiation. This is thought to deliver a more lethal dose of radiation to the tumor and is more convenient with treatment being completed within 2-3 weeks compared to the typical 7-8 week course of conventional radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed, by biopsy or cytology, non-small cell lung carcinoma diagnosed within 3 months prior to study enrollment.
* T1, N0, M0 or T2, N0, M0. (AJCC Lung 7th Edition)
* At least 18 years old at the time of consent.
* Adequate bone marrow function.
* Medically inoperable. Medically operable candidates are allowed if they refuse surgical resection.
* If the patient has a large pleural effusion, it must be biopsy negative.

Exclusion Criteria:

* Evidence of distant metastasis (M1) and/or nodal involvement (N1, N2, N3).
* Synchronous primary.
* T2 tumors > 5 cm; T3, T4 primary tumor.
* Previous radiotherapy for lung cancer.
* Concomitant local, regional, and/or systemic therapy during radiotherapy.
* Active systemic, pulmonary, and/or pericardial infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Confirm Grade 3 or higher toxicity rate of hypoIGRT proton therapy in patients with stage I non-small cell lung cancer. | 1 year after the end of radiation therapy

SECONDARY OUTCOMES:
Collect and analyze outcome data on tumor control and survival | When each patient has been followed for a minimum of 12 months to a maximum of 5 years
Assess differences in dosimetric values compared with photons for lung, heart, esophagus, spinal cord, skin and brachial plexus | When each patient has been followed for a minimum of 12 months to a maximum of 5 years
Assess changes in quality of life before and after treatment | Before treatment and then when each patient has been followed for a minimum of 12 months to a maxiumum of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Romaine C Nichols, MD, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Murray T, Thun MJ. Cancer statistics, 2008. CA Cancer J Clin. 2008 Mar-Apr;58(2):71-96. doi: 10.3322/CA.2007.0010. Epub 2008 Feb 20. PMID 18287387
- [Background] al-Kattan K, Sepsas E, Fountain SW, Townsend ER. Disease recurrence after resection for stage I lung cancer. Eur J Cardiothorac Surg. 1997 Sep;12(3):380-4. doi: 10.1016/s1010-7940(97)00198-x. PMID 9332915
- [Background] Suzuki K, Nagai K, Yoshida J, Moriyama E, Nishimura M, Takahashi K, Nishiwaki Y. Prognostic factors in clinical stage I non-small cell lung cancer. Ann Thorac Surg. 1999 Apr;67(4):927-32. doi: 10.1016/s0003-4975(99)00140-x. PMID 10320230
- [Background] van Rens MT, de la Riviere AB, Elbers HR, van Den Bosch JM. Prognostic assessment of 2,361 patients who underwent pulmonary resection for non-small cell lung cancer, stage I, II, and IIIA. Chest. 2000 Feb;117(2):374-9. doi: 10.1378/chest.117.2.374. PMID 10669677
- [Background] Dosoretz DE, Galmarini D, Rubenstein JH, Katin MJ, Blitzer PH, Salenius SA, Dosani RA, Rashid M, Mestas G, Hannan SE, et al. Local control in medically inoperable lung cancer: an analysis of its importance in outcome and factors determining the probability of tumor eradication. Int J Radiat Oncol Biol Phys. 1993 Oct 20;27(3):507-16. doi: 10.1016/0360-3016(93)90373-4. PMID 8226142
- [Background] Dosoretz DE, Katin MJ, Blitzer PH, Rubenstein JH, Salenius S, Rashid M, Dosani RA, Mestas G, Siegel AD, Chadha TT, et al. Radiation therapy in the management of medically inoperable carcinoma of the lung: results and implications for future treatment strategies. Int J Radiat Oncol Biol Phys. 1992;24(1):3-9. doi: 10.1016/0360-3016(92)91013-d. PMID 1324899
- [Background] Gauden S, Ramsay J, Tripcony L. The curative treatment by radiotherapy alone of stage I non-small cell carcinoma of the lung. Chest. 1995 Nov;108(5):1278-82. doi: 10.1378/chest.108.5.1278. PMID 7587429
- [Background] Baumann P, Nyman J, Lax I, Friesland S, Hoyer M, Rehn Ericsson S, Johansson KA, Ekberg L, Morhed E, Paludan M, Wittgren L, Blomgren H, Lewensohn R. Factors important for efficacy of stereotactic body radiotherapy of medically inoperable stage I lung cancer. A retrospective analysis of patients treated in the Nordic countries. Acta Oncol. 2006;45(7):787-95. doi: 10.1080/02841860600904862. PMID 16982541
- [Background] Fritz P, Kraus HJ, Blaschke T, Muhlnickel W, Strauch K, Engel-Riedel W, Chemaissani A, Stoelben E. Stereotactic, high single-dose irradiation of stage I non-small cell lung cancer (NSCLC) using four-dimensional CT scans for treatment planning. Lung Cancer. 2008 May;60(2):193-9. doi: 10.1016/j.lungcan.2007.10.005. Epub 2007 Nov 28. PMID 18045732
- [Background] Lagerwaard FJ, Haasbeek CJ, Smit EF, Slotman BJ, Senan S. Outcomes of risk-adapted fractionated stereotactic radiotherapy for stage I non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2008 Mar 1;70(3):685-92. doi: 10.1016/j.ijrobp.2007.10.053. Epub 2007 Dec 31. PMID 18164849
- [Background] Onishi H, Shirato H, Nagata Y, Hiraoka M, Fujino M, Gomi K, Niibe Y, Karasawa K, Hayakawa K, Takai Y, Kimura T, Takeda A, Ouchi A, Hareyama M, Kokubo M, Hara R, Itami J, Yamada K, Araki T. Hypofractionated stereotactic radiotherapy (HypoFXSRT) for stage I non-small cell lung cancer: updated results of 257 patients in a Japanese multi-institutional study. J Thorac Oncol. 2007 Jul;2(7 Suppl 3):S94-100. doi: 10.1097/JTO.0b013e318074de34. PMID 17603311
- [Background] Timmerman R, McGarry R, Yiannoutsos C, Papiez L, Tudor K, DeLuca J, Ewing M, Abdulrahman R, DesRosiers C, Williams M, Fletcher J. Excessive toxicity when treating central tumors in a phase II study of stereotactic body radiation therapy for medically inoperable early-stage lung cancer. J Clin Oncol. 2006 Oct 20;24(30):4833-9. doi: 10.1200/JCO.2006.07.5937. PMID 17050868
- [Background] Xia T, Li H, Sun Q, Wang Y, Fan N, Yu Y, Li P, Chang JY. Promising clinical outcome of stereotactic body radiation therapy for patients with inoperable Stage I/II non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2006 Sep 1;66(1):117-25. doi: 10.1016/j.ijrobp.2006.04.013. Epub 2006 Jun 9. PMID 16765528
- [Background] Hof H, Muenter M, Oetzel D, Hoess A, Debus J, Herfarth K. Stereotactic single-dose radiotherapy (radiosurgery) of early stage nonsmall-cell lung cancer (NSCLC). Cancer. 2007 Jul 1;110(1):148-55. doi: 10.1002/cncr.22763. PMID 17516437
- [Background] Zimmermann FB, Geinitz H, Schill S, Thamm R, Nieder C, Schratzenstaller U, Molls M. Stereotactic hypofractionated radiotherapy in stage I (T1-2 N0 M0) non-small-cell lung cancer (NSCLC). Acta Oncol. 2006;45(7):796-801. doi: 10.1080/02841860600913210. PMID 16982542
- [Background] Yamashita H, Nakagawa K, Nakamura N, Koyanagi H, Tago M, Igaki H, Shiraishi K, Sasano N, Ohtomo K. Exceptionally high incidence of symptomatic grade 2-5 radiation pneumonitis after stereotactic radiation therapy for lung tumors. Radiat Oncol. 2007 Jun 7;2:21. doi: 10.1186/1748-717X-2-21. PMID 17553175
- [Background] Onimaru R, Shirato H, Shimizu S, Kitamura K, Xu B, Fukumoto S, Chang TC, Fujita K, Oita M, Miyasaka K, Nishimura M, Dosaka-Akita H. Tolerance of organs at risk in small-volume, hypofractionated, image-guided radiotherapy for primary and metastatic lung cancers. Int J Radiat Oncol Biol Phys. 2003 May 1;56(1):126-35. doi: 10.1016/s0360-3016(03)00095-6. PMID 12694831
- [Background] Georg D, Hillbrand M, Stock M, Dieckmann K, Potter R. Can protons improve SBRT for lung lesions? Dosimetric considerations. Radiother Oncol. 2008 Sep;88(3):368-75. doi: 10.1016/j.radonc.2008.03.007. Epub 2008 Apr 9. PMID 18405986
- [Background] Bush DA, Slater JD, Shin BB, Cheek G, Miller DW, Slater JM. Hypofractionated proton beam radiotherapy for stage I lung cancer. Chest. 2004 Oct;126(4):1198-203. doi: 10.1378/chest.126.4.1198. PMID 15486383
- [Background] Miyamoto T, Baba M, Sugane T, Nakajima M, Yashiro T, Kagei K, Hirasawa N, Sugawara T, Yamamoto N, Koto M, Ezawa H, Kadono K, Tsujii H, Mizoe JE, Yoshikawa K, Kandatsu S, Fujisawa T; Working Group for Lung Cancer. Carbon ion radiotherapy for stage I non-small cell lung cancer using a regimen of four fractions during 1 week. J Thorac Oncol. 2007 Oct;2(10):916-26. doi: 10.1097/JTO.0b013e3181560a68. PMID 17909354
- [Background] Lagerwaard FJ et al Quality of life after stereotactic radiotherapy for medically inoperable stage I lung cancer. International Journal of Radiation Oncology, Biology, Physics IJROBP 2006 Nov1;66(3): S133-S134
- [Background] Brown J, Thorpe H, Napp V, Fairlamb DJ, Gower NH, Milroy R, Parmar MK, Rudd RM, Spiro SG, Stephens RJ, Waller D, West P, Peake MD. Assessment of quality of life in the supportive care setting of the big lung trial in non-small-cell lung cancer. J Clin Oncol. 2005 Oct 20;23(30):7417-27. doi: 10.1200/JCO.2005.09.158. Epub 2005 Sep 12. PMID 16157935
- [Background] Li WW, Lee TW, Lam SS, Ng CS, Sihoe AD, Wan IY, Yim AP. Quality of life following lung cancer resection: video-assisted thoracic surgery vs thoracotomy. Chest. 2002 Aug;122(2):584-9. doi: 10.1378/chest.122.2.584. PMID 12171836